CLINICAL TRIAL: NCT03669536
Title: Determinants of Cognitive Impairment Among Geriatrics in an Indonesian Old Age Home
Brief Title: Determinants of Cognitive Impairment Among Geriatrics
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tarumanagara University (Other)
Collaborators: Hana Old Age Home (Unknown)
Responsible Party: Principal Investigator, Anthony Paulo Sunjaya, Principal Investigator, Tarumanagara University
Other Study IDs: APS007
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Impairment; Dementia; Hearing Impairment; Vision Impairment and Blindness; Diabetes; Dyslipidemias; Obesity; Central Obesity; Mobility Limitation; Osteoarthritis; Hypertension; Depression
Keywords: cognitive impairment; dementia; geriatrics
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Hearing Loss; Vision Disorders; Blindness; Diabetes Mellitus; Dyslipidemias; Obesity; Obesity, Abdominal; Mobility Limitation; Osteoarthritis; Hypertension; Depression

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the determinants of cognitive impairment among Indonesian geriatrics in an Old Age Home.

DETAILED DESCRIPTION:
Elderly patients (≥ 60 years of age) are enrolled in this study. The inclusion criteria are patients which have consented to take part in the study.

Data such as age, ethnic, education, BMI, waist and hip circumference, blood pressure, hearing impairment, vision impairment, depression, sleep disorder, mobility, hemoglobin levels, glycemic and lipid profile, as well as comorbidities and drugs used were collected from the patients' medical records, laboratory tests and through examination by trained examiners.

Cognition was determined through a combination of several psychiatric examinations using validated instruments namely - MiniCog, Clock Drawing Test, Three Word Recall, Alzheimer's Disease-8 Indonesia (AD-8 INA) Questionnaire and Short Portable Mental Status Questionnaire (SPMSQ).

ELIGIBILITY:
Inclusion Criteria:

* Must be classified as geriatric according to Indonesian Laws (≥ 60 years of age).
* Consented to participate in this study.

Exclusion Criteria:

* Uncooperative.
* Incomplete records.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly patients (≥ 60 years of age) currently under the care of an Indonesian Old Age Home.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
MiniCog | Through study completion, an average of 6 months
  Based on psychiatric examination using the Indonesian MiniCog Questionnaire to determine patient's cognitive status. A MiniCog result below 5 implies mild cognitive impairment, while a result below 3 implies dementia.
Clock Drawing Test (CDT) | Through study completion, an average of 6 months
  Based on psychiatric examination using the Indonesian Clock Drawing Test to determine patient's cognitive status. A Clock Drawing Test score below 4 implies mild cognitive impairment.
Three Word Recall | Through study completion, an average of 6 months
  Based on psychiatric examination using the Indonesian Three Word Recall Test to determine patient's cognitive status with resulting score from 0-3. Zero means no words can be recalled by the patient.
Alzheimer Disease-8 Indonesia Questionnaire (AD-8 INA) | Through study completion, an average of 6 months
  Based on interviews with caretakers using the AD-8 INA Questionnaire to determine patient's cognitive status. An AD-8 INA score of 2 or more implies mild cognitive impairment.
Short Portable Mental Status Questionnaire (SPMSQ) | Through study completion, an average of 6 months
  Based on psychiatric examination using the Indonesian SPMSQ to determine patient's cognitive status. An SPMSQ test in which the patient demonstrated more than 3 mistakes implies mild cognitive impairment, whereas a mistake of greater than 8 implies dementia.

OTHER OUTCOMES:
Hearing Impairment | Through study completion, an average of 6 months
  Based on physical examination using the Whispered Sound Test from 6 meters and tuning fork test as well as history of hearing impairment from medical records.
Vision Impairment | Through study completion, an average of 6 months
  Based on physical examination using the Snellen Chart and history of vision impairment from medical records.
Diabetes | Through study completion, an average of 6 months
  Based on glycemic profile results and history of diabetes from medical records. Patients are classified as diabetic in accordance to the Indonesian Society of Endocrinology and American Diabetic Association criteria.
Mobility | Through study completion, an average of 6 months
  Based on physical examination, Indonesian Validated Lequesne Index, Barthel Acitivities of Daily Living (ADL), Instrumental ADL and history of arthritis or other pathologies affecting mobility from medical records.
Depression | Through study completion, an average of 6 months
  Based on psychiatric examination, Indonesian Validated Geriatric Depression Scale and Medical Records. A score of 5-9 implies a likelihood of depression, while a score of greater than 10 implies depression.
Sleep Disorder | Through study completion, an average of 6 months
  Based on psychiatric examination, Indonesian Validated Insomnia Severity Index and Medical Records. A score of 8-14 implies mild insomnia, 15-21 intermediate insomnia and 22-28 severe insomnia.
Hypertension | Through study completion, an average of 6 months
  Based on blood pressure results and history of hypertension from medical records.
Dyslipidemia | Through study completion, an average of 6 months
  Based on lipid profile results and history of dyslipidemia from medical records.
Anemia | Through study completion, an average of 6 months
  Based on hemoglobin results.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sunjaya, Principal Investigator — Tarumanagara University
Locations (1):
- Hana Old Age Home, Tangerang, Banten, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided